CLINICAL TRIAL: NCT06939777
Title: A Randomized, Double-Blind, Controlled, Phase I/II Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of SNA02-48 Injection in Chinese Adult Participants
Brief Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of SNA02-48 Injection in Chinese Adult Participants
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sinovac Life Sciences Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Sinovac Biotech Co., Ltd (Industry)
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PRO-SNA02-48-1001
Record Dates: First submitted 2025-04-15; First posted 2025-04-23 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Tetanus
MeSH Terms: conditions — Tetanus | interventions — Tetanus Toxoid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (12):
- Cohort 1:low-dose SNA02-48/placebo (Phase I) (Experimental): Participants will be randomly assigned to receive either low-dose SNA02-48 or placebo.
  Interventions: Biological: SNA02-48; Biological: Placebo
- Cohort 2: medium-dose SNA02-48/placebo (Phase I) (Experimental): Participants will be randomly assigned to receive either medium-dose SNA02-48 or placebo.
  Interventions: Biological: SNA02-48; Biological: Placebo
- Cohort 3: high-dose SNA02-48/placebo (Phase I) (Experimental): Participants will be randomly assigned to receive either high-dose SNA02-48 or placebo.
  Interventions: Biological: SNA02-48; Biological: Placebo
- Group A :low-dose SNA02-48 + placebo (Phase II) (Experimental): Participants will receive a single intramuscular (IM) gluteal injection of low-dose SNA02-48 and a single IM deltoid injection of placebo
  Interventions: Biological: SNA02-48; Biological: Placebo
- Group B : medium-dose SNA02-48 + placebo (Phase II) (Experimental): Participants will receive a single IM gluteal injection of medium-dose SNA02-48 and a single IM deltoid injection of placebo
  Interventions: Biological: SNA02-48; Biological: Placebo
- Group C : high-dose SNA02-48 + placebo (Phase II) (Experimental): Participants will receive a single IM gluteal injection of high-dose SNA02-48 and a single IM deltoid injection of placebo
  Interventions: Biological: SNA02-48; Biological: Placebo
- Group D : low-dose SNA02-48 + Tetanus Toxoid (Phase II) (Experimental): Participants will receive a single IM gluteal injection of low-dose SNA02-48 and a single IM deltoid injection of Tetanus Toxoid（TT）
  Interventions: Biological: SNA02-48; Biological: Tetanus Toxoid
- Group E : medium-dose SNA02-48 + Tetanus Toxoid (Phase II) (Experimental): Participants will receive a single IM gluteal injection of medium-dose SNA02-48 and a single IM deltoid injection of Tetanus Toxoid（TT）
  Interventions: Biological: SNA02-48; Biological: Tetanus Toxoid
- Group F : high-dose SNA02-48 + Tetanus Toxoid (Phase II) (Experimental): Participants will receive a single IM gluteal injection of high-dose SNA02-48 and a single IM deltoid injection of Tetanus Toxoid（TT）
  Interventions: Biological: SNA02-48; Biological: Tetanus Toxoid
- Group G : placebo + Tetanus Toxoid (Phase II) (Placebo Comparator): Participants will receive a single IM gluteal injection of placebo and a single IM deltoid injection of Tetanus Toxoid（TT）
  Interventions: Biological: Placebo; Biological: Tetanus Toxoid
- Group H : Human tetanus immunoglobulin(HTIG) + placebo (Phase II) (Active Comparator): Participants will receive a single IM gluteal injection of Human tetanus immunoglobulin(HTIG) and a single IM deltoid injection of placebo
  Interventions: Biological: Placebo; Biological: HTIG
- Group I : Human tetanus immunoglobulin(HTIG) + Tetanus Toxoid（TT） (Phase II) (Active Comparator): Participants will receive a single IM gluteal injection of Human tetanus immunoglobulin(HTIG) and a single IM deltoid injection of Tetanus Toxoid（TT）
  Interventions: Biological: HTIG; Biological: Tetanus Toxoid

INTERVENTIONS:
Biological: SNA02-48 — intramuscular injection
  Arms: Cohort 1:low-dose SNA02-48/placebo (Phase I); Cohort 2: medium-dose SNA02-48/placebo (Phase I); Cohort 3: high-dose SNA02-48/placebo (Phase I); Group A :low-dose SNA02-48 + placebo (Phase II); Group B : medium-dose SNA02-48 + placebo (Phase II); Group C : high-dose SNA02-48 + placebo (Phase II); Group D : low-dose SNA02-48 + Tetanus Toxoid (Phase II); Group E : medium-dose SNA02-48 + Tetanus Toxoid (Phase II); Group F : high-dose SNA02-48 + Tetanus Toxoid (Phase II)
Biological: Placebo — intramuscular injection
  Arms: Cohort 1:low-dose SNA02-48/placebo (Phase I); Cohort 2: medium-dose SNA02-48/placebo (Phase I); Cohort 3: high-dose SNA02-48/placebo (Phase I); Group A :low-dose SNA02-48 + placebo (Phase II); Group B : medium-dose SNA02-48 + placebo (Phase II); Group C : high-dose SNA02-48 + placebo (Phase II); Group G : placebo + Tetanus Toxoid (Phase II); Group H : Human tetanus immunoglobulin(HTIG) + placebo (Phase II)
Biological: HTIG — intramuscular injection
  Arms: Group H : Human tetanus immunoglobulin(HTIG) + placebo (Phase II); Group I : Human tetanus immunoglobulin(HTIG) + Tetanus Toxoid（TT） (Phase II)
Biological: Tetanus Toxoid — intramuscular injection
  Arms: Group D : low-dose SNA02-48 + Tetanus Toxoid (Phase II); Group E : medium-dose SNA02-48 + Tetanus Toxoid (Phase II); Group F : high-dose SNA02-48 + Tetanus Toxoid (Phase II); Group G : placebo + Tetanus Toxoid (Phase II); Group I : Human tetanus immunoglobulin(HTIG) + Tetanus Toxoid（TT） (Phase II)

SUMMARY:
To evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics of the full human anti-tetanus toxin monoclonal antibody SNA02-48 injection and compare the Tetanus-antibody levels and safety of SNA02-48 with human tetanus immunoglobulin (HTIG) in Chinese adult participants.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo/active-controlled phase I/II study to evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics of SNA02-48 Injection in Chinese adult participants.

In the phase I portion of the study, 30 adult participants will be sequentially enrolled into three cohorts. Each participant will receive a single intramuscular (IM) dose of either SNA02-48 or placebo, depending on the cohort to which they are assigned. The phase I part will last for 105 days following the assessments of safety, PK, PD and ADA.

In the phase II portion of the study, 225 adult participants will be enrolled and randomly assigned to nine groups.The phase II part will last for 105 days following the assessments of safety, PK, PD and ADA.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 18-59 years of age；
2. Participants have the ability to understand and agree to sign the informed consent form；
3. Male participants with a weight of≥50.0kg; Female participants with a weight of ≥ 45.0kg and the weight of both men and women≤90 kg, 18.5 kg/m2≤BMI < 24.0 kg/m2;
4. Participants of childbearing potential and their sexual partners voluntarily adopt effective contraceptive measures from the date of signing the informed consent form until 6 months after the administration of the investigational drug, and have no plans to donate sperm or ova during this period.

Exclusion Criteria:

1. Previous history of tetanus infection;
2. Has received tetanus vaccines or vaccines containing tetanus toxoid antigen (DTP, DT, meningococcal conjugate vaccine, etc.) within the last 10 years, or has received a tetanus immunoglobulin or tetanus antitoxin within the previous 6 months;
3. Participants with positive tetanus antibody IgG test results during the screening period；
4. Participants who are known to be allergic to experimental drugs (including excipients, HTIG, and other therapeutic monoclonal antibodies), or who suffer from severe allergic diseases, may damage the safety of the participants by the judgment of the investigator;
5. Positive for hepatitis B surface antigen (HBsAg), hepatitis C antibody (HCV Ab), HIV antibody (HIV Ab), or Treponema pallidum antibody (TP Ab);
6. Physical examinations, vital signs, electrocardiograms (ECGs), laboratory tests, or other test results during the screening or baseline period that are judged by the investigator to be abnormal and clinically significant;
7. Participants with uncontrolled chronic or severe disease history, including but not limited to cardiovascular disease, hematological system disease, hepatobiliary or renal diseases, gastrointestinal diseases, respiratory disease, malignant tumor, history of major organ transplantation, which may affect the pharmacokinetic profiles or safety evaluation of the investigational drug as determined by the investigator;
8. Autoimmune diseases or immunodeficiency disorders (including but not limited to systemic lupus erythematosus (SLE), ankylosing spondylitis (AS), autoimmune thyroid diseases (AITD), asplenia, functional asplenia, or human immunodeficiency virus infection (HIV));
9. Participants with coagulation dysfunction that is abnormal and clinically significant as determined by the investigator (e.g., coagulation factor deficiency, platelet abnormalities);
10. Current or past history of severe neurological disorders (including but not limited to epilepsy, convulsions, or seizures) or psychiatric disorders, or a family history of psychiatric disorders;
11. Have a history of drug abuse or dependence or recreational drug use within 2 years prior to screening, or have a positive urine drug abuse screening before enrollment;
12. Participants who have received immunosuppressants or other immunomodulatory therapies (e.g., prednisone≥20 mg/day or equivalent) for≥14 days within the 6 months, cytotoxic therapy, or plan to receive such treatments during the trial period;
13. Participants who have received immune globulin or other blood products within the 6 months, or plan to receive such treatments during the trial period;
14. Participants who have donated >400 ml of blood or experienced significant blood loss >400 ml within 3 months prior to drug administration, or donated plasma or platelets within 1 month prior to drug administration;
15. Participants who have participated in other drug or medical device clinical trials within 3 months prior to screening, or plan to participate in other clinical trials during the trial period;
16. Participants who have smoked≥5 cigarettes per day within 3 months prior to screening;
17. Participants who have consumed >14 alcohol units per week within 3 months prior to screening (1 alcohol unit = 14 grams of pure alcohol = 360 ml beer, 150 ml wine, or 45 ml distilled spirits/liquor);
18. Acute diseases, acute exacerbation of chronic diseases or surgical history within 4 weeks prior to screening;
19. Receipt of live attenuated vaccines within 4 weeks prior to screening or subunit/inactivated vaccines (or other vaccine types) within 7 days prior to screening;
20. Receipt of any prescription medications, over-the-counter (OTC) medications supplements, or functional vitamins within 14 days prior to screening;
21. Participants who have consumed special diets (e.g., grapefruit, etc.) or engaged in strenuous exercise, or have other factors affecting drug absorption, distribution, metabolism, or excretion within 14 days prior to screening;
22. Women in pregnancy or lactation or those with a positive pregnancy test;
23. Participants who have consumed any caffeine-containing or tea within 24 hours prior to investigational drug administration;
24. Ear temperature during the screening or baseline period is> 37.6℃;
25. Skin lesions (including inflammation, ulcers, rashes, or scars) at the target injection site that may interfere with drug administration or observation of local reactions;
26. According to the investigator's judgment, the subject has any other factors that are not suitable for participating in the clinical trial.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 255 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse reactions | Up to 105 days
The increase in serum tetanus antibody levels from baseline at 12 hours post-administration | 12 hours after administration

SECONDARY OUTCOMES:
Time of maximum plasma concentration (Tmax) | Up to 105 days
Peak plasma concentration(Cmax) | Up to 105 days
Terminal half-life (T1/2) | Up to 105 days
clearance(CL) | Up to 105 days
Apparent Volume of Distribution(Vd) | Up to 105 days
Area under the plasma concentration time curve (AUC) | Up to 105 days
Terminal Elimination Rate Constant(λz) | Up to 105 days
Mean Residence Time (MRT) | Up to 105 days
Serum tetanus antibody level | Up to 105 days
Positive rate of serum tetanus antibody | Up to 105 days
The increase in serum tetanus antibody levels from baseline after administration | Up to 105 days
Incidence of anti-drug antibody (ADA) and neutralizing antibody (Nab) | Up to 105 days

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Hospital of Anhui Medical University, Hefei, Anhui, China